CLINICAL TRIAL: NCT04308655
Title: Obstetric Pain Management for Women With Opioid Use Disorder: A Longitudinal, Qualitative Mixed-methods Evaluation of Patients and Provider Perspectives
Brief Title: Obstetric Pain Management for Women With Opioid Use Disorder (QUEST)
Acronym: QUEST
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Grace Lim, MD, MS, Primary Investigator, University of Pittsburgh
Other Study IDs: STUDY20010041
Record Dates: First submitted 2020-03-06; First posted 2020-03-16 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Interviews as Topic; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient participants: This cohort will include pregnant patients with a history of opiate use disorder (OUD) who will be followed from the third trimester of pregnancy until five days postpartum.
  Interventions: Other: Interview; Other: Surveys
- Provider participants: This cohort will include clinicians who provide care for pregnant patients with OUD. Providers will be interviewed and will complete one survey cross-sectionally.
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — Semi-structured interviews
Other: Surveys — Validated surveys on pain, fear, anxiety, depression, beliefs
  Groups: Patient participants

SUMMARY:
This is a mixed methods longitudinal observational study to assess patient and provider perspectives on pain and pain management among pregnant women with opiate use disorder (OUD). The findings from this study will inform patient-centered approaches to pain management. Themes surrounding mothers' pain/recovery experiences that correlate with quantified pain and analgesia endpoints will be identified. Findings will also shape an appropriate patient-centered research agenda for obstetric pain management in patients with OUD.

DETAILED DESCRIPTION:
A fine understanding of the attitudes and beliefs about pain and its management for patients with opioid use disorder is currently lacking. These psychological aspects of pain and analgesia are expected to have significant effects on nociception, pain experience, analgesic efficacy, and opioid requirements and its subsequent risks for relapse/treatment noncompliance. There is also have little understanding of provider-held attitudes and beliefs which can influence pain and its treatment for this population.

The findings from this study will inform patient-centered approaches to pain management for obstetric patients with OUD. They will also shape an appropriate patient-centered research agenda for obstetric pain management in patients with OUD. This work will find new patient-centered endpoints for this special population that may be currently overlooked with existing standard pain assessments.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who are 18 years of age or older
* History of opioid use disorder, on medication assisted therapy
* Currently in their third trimester

Exclusion Criteria:

* Unable to participate in informed consent discussions
* Unable to give informed consent for any reason
* Not fluent in English (surveys are validated in English language)
* Unable to participate fully in all study procedures for any reason

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will enroll pregnant adults with opiate use disorder (on medication assisted therapy) who are currently in their third trimester.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2020-03-06 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Themes surrounding mothers' pain/recover experience | Through study completion, an average of 6 weeks (from enrollment through labor and delivery)
  The endpoint of this mixed-methods investigation is to identify themes surrounding mothers' pain/recovery experiences that correlate with quantified pain and analgesic needs. Endpoint will take the form of words/terms, phrases, or sentences. Identification of these terms, phases, or sentences are not identified a priori in this qualitative investigation.

CONTACTS AND LOCATIONS:
Overall Officials: Grace Lim, MD MS, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Magee Womens Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No